CLINICAL TRIAL: NCT04559997
Title: 6-year Follow-up Study of the Effectiveness of Neurorehabilitation Treatment in a Patient With Parkinson's Disease
Brief Title: A 6-year Follow-up Study of the Effect of Neurorehabilitation Training in Patients With Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Somogy Megyei Kaposi Mór Teaching Hospital (Other)
Responsible Party: Principal Investigator, Tollár József, Dr. József Tollár, 7400 Kaposvár, Tallián Gy. u 20-32, Somogy Megyei Kaposi Mór Teaching Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IKEB2020/05
Record Dates: First submitted 2020-09-10; First posted 2020-09-23 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Follow up; Parkinson Disease; Rehabilitation
Keywords: balance; Posturograpy
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Exercise+FU (Experimental): Parkinson's group takes part in a treadmill treatment that takes place 3 times a week for 6 years.
  Interventions: Other: Exercise+FU
- Exercise (Active Comparator): After 3 weeks of intensive treatment, no special exercises are performed as a control.
  Interventions: Other: Active Comparator group Exercise
- Controll (No Intervention): No intervention.

INTERVENTIONS:
Other: Exercise+FU — 6 years intervention, administered daily, targeted postural instability, balance and mobility using at-limit intensity sensorimotor and visuomotor agility training
  Arms: Exercise+FU
Other: Active Comparator group Exercise — After 3 weeks of intensive therapy, we withdrew treatment and monitored their condition for 6 years and received only hospital base treatment
  Arms: Exercise

SUMMARY:
Individualization of exercise is recommended but rarely performed in patients with Parkinson's disease (PD). Unusually High Intensity and Individual Sensor Motor with Visuomotor Mobility Trainer The clinical symptoms, mobility and posture of PD patients. After 3 weeks of intensive treatment, treated patients and the control group were subjected to a two-year observation. Objectives: The effect of the unusually highly intense and strictly individualized sensomotor and visuomotor agility program was determined for the clinical symptoms, mobility and stability of non-demented PD patients with a two-year follow-up. Detection and comparison of results of patients undergoing biphasic maintenance with the results of intensively treated patients and the control group. Patients were recalled every 3 months after the first intensive examination and one year after a one-year control. The results of the active group were continuously compared with the results of the passive and control groups, thus determining the effectiveness of our treatment and the deterioration of the other groups in life-quality. The treated groups will be divided into two. One Parkinson's group takes part in a treadmill treatment that takes place 3 times a week for 6 years. The other group does not undergo a special series of exercises after 3 weeks of intensive therapy. Main outcome measures: Movement disorder Society Unified Parkinson Disease Rating Scale, Motor Experiences of Daily Living, a measure sensitive to changes in a broad spectrum of PD symptoms. In group time, repeated measurements of variance analysis were compared to MDS-UPDRS M-EDL, Beck Depression Score, PDQ-39, EQ5D VAS, Schwab & England Scale for Parkinson's Disease. The TUG test and 12 static posturographic measurements are compared and compared to the healthy group as a standard. An at-limit and individualized sensorimotor and visuomotor agility exercise program vs. standard care, will improve non-demeted, stage 2-3 PD patient's clinical symptoms, mobility, and postural stability by functionally meaningful margins. As a long-term solution, a follow-up treatment can slow down the progression of clinical symtoms.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's disease
* Hoenh Yahr scale of 2-3
* Instability problem

Exclusion Criteria:

* Severe heart problems
* Severe demeanor
* Alcoholism
* Drug problems

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2014-09-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
EQ5D-5L | 6 years long
  Questionnaire
posturography | 6 year-long
  body sway, Objective measurement of holding instability
Timed up and Go test | 6 year-long
  Measuring the speed of walking

CONTACTS AND LOCATIONS:
Locations (1):
- Somogy Megyei Kaposi Mór Oktató Kórház, Kaposvár, Somogy County, Hungary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/?term=parkinson+rehabilitation